CLINICAL TRIAL: NCT02638714
Title: Treatment of Optic Neuropathies Using Autologous Bone-Marrow Derived Clusters of Differentiation (CD) 34+, 133+, and 271+ Stem Cells: A Pilot Study
Brief Title: Treatment of Optic Neuropathies Using Autologous Bone Marrow-Derived Stem Cells
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stem Cells Arabia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCA-ON1
Record Dates: First submitted 2015-12-07; First posted 2015-12-23 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Optic Neuropathy
Keywords: Optic Neuropathies; Stem Cell Therapy
MeSH Terms: conditions — Optic Nerve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cells (Experimental): Intervention: Transplantation of autologous purified stem cells
  Interventions: Biological: Stem Cells

INTERVENTIONS:
Biological: Stem Cells — Intervention: Transplantation of autologous purified stem cells

SUMMARY:
A single arm, single center trial to assess the safety and efficacy of restoring function in damaged optic nerves using autologous purified populations of bone-marrow derived stem cells (BM-SCs) through a 24 month follow up period.

DETAILED DESCRIPTION:
Optic nerve atrophy (ONA) is a condition defined as a damage to the optic nerve that harmfully affects central and peripheral vision. ONA may occur as a result of optic neuritis, compression by tumors or aneurysms, toxic and nutritional neuropathies, trauma, or as a secondary complication to other systemic diseases such as diabetes. Symptoms of ONA vary diversely, but mainly include blurred vision and a reduction in optic sharpness and color visualization. ONA is irreversible process, and current medical strategies focus on finding the underlying cause, and trying to prevent further vision loss and protect the other healthy eye. This is a Single arm, Single Center trial to assess the safety and efficacy of purified adult autologous bone marrow derived CD34+, CD133+, and CD271+ stem cells through a 24 month follow-up period. The combination of these three cell types was based on their diverse potentialities to differentiate into specific functional cell types to regenerate damaged optic nerves and supporting issues and vasculature, and the availability of clinical-grade purification system (CliniMACS) and Microbeads to purify the target cell populations in clinically-approved methods. Anticipated outcomes of this study are defined in an overall improvement of vision, restoration of functions to damaged optic nerves, and improvement in quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient should suffer from Optic Nerve Atrophy diseases like diabetic retinopathy and retinal pigmentation.
* Age in between 18-55 years old
* Willingness to undergo bone marrow derived autologous cell therapy.
* Ability to comprehend the explained protocol
* Ability and willingness to regularly visit to hospital for protocol and follow up

Exclusion Criteria:

* Patients with preexisting or current systemic disease such as lung, liver, gastrointestinal, cardiac, immunodeficiency, syphilis, or clinically relevant polyneuropathies.
* History of life threatening allergic or immune- mediated reaction

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-04; Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in degeneration of the optic nerve using the visual field assessment with the Humphrey automated and Goldmann manual perimeters | 24 months

SECONDARY OUTCOMES:
improvement in visual function using the documentation of visual acuity using the Snellen chart | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Adeeb AlZoubi, PhD, Principal Investigator
Locations (1):
- Stem Cells of Arabia, Amman, Jordan